CLINICAL TRIAL: NCT00029653
Title: The Effect of Transcranial Magnetic Stimulation on Free Will
Brief Title: Effect of Transcranial Magnetic Stimulation on Free Will
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020101; 02-N-0101
Record Dates: First submitted 2002-01-16; First posted 2002-01-17 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Healthy
Keywords: Frontal Lobe; Reaction Time; Movement Preparation; Motor Threshold; Transcranial Magnetic Stimulation; Motor Cortex; Healthy Volunteer; Normal Control; HV

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) to investigate how the brain controls movement by sending messages to the spinal cord and muscles.

Healthy normal volunteers 21 years of age or older may participate in this study.

They must have no medical, neurological or psychiatric illnesses nor have been taking medications that affect nervous system function.

Participants will undergo transcranial magnetic stimulation. For this procedure, an insulated wire coil is placed on the scalp or skin. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. If the coil is placed over a nerve or area of the brain that controls muscles, it may cause a muscle twitch, possibly strong enough to move the limb. In other cases, the subject may have a feeling of movement or feel a tingling sensation in a limb. Stimulation over the muscles on the side of the head may cause some discomfort in that area or twitching of the jaw.

During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The electrical activity of the muscles activated by the stimulation will be recorded using metal electrodes taped to the skin over the muscle. In most cases, the study takes less than 3 hours.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the influence of transcranial magnetic stimulation (TMS) on free will to select movement. There have been debates that most of human voluntary movements are reflexive rather than volitional in nature, although most people feel that their movements are freely chosen. This issue is illuminated by previous TMS studies showing external bias of freely chosen movements by TMS. Recently, we tried to confirm these observations using a more reliable method with subthreshold TMS, but failed. Thus, in this study, we are planning to use suprathreshold TMS to test whether this type of stimulation on different motor areas influences free selection of movements or not.

ELIGIBILITY:
Normal adult volunteers who are 21 years or older will be eligible.

Volunteers who have either any medico-surgical, neurological and psychiatric illnesses, who have been taking any medication with potential influence on nervous system function, who have a pacemaker, an implanted medical pump, a metal plate or a metal object in the skull or eye (for example, after brain surgery), or who have a history of seizure disorder, will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2002-01; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Prochazka A, Clarac F, Loeb GE, Rothwell JC, Wolpaw JR. What do reflex and voluntary mean? Modern views on an ancient debate. Exp Brain Res. 2000 Feb;130(4):417-32. doi: 10.1007/s002219900250. PMID 10717785
- [Background] Ammon K, Gandevia SC. Transcranial magnetic stimulation can influence the selection of motor programmes. J Neurol Neurosurg Psychiatry. 1990 Aug;53(8):705-7. doi: 10.1136/jnnp.53.8.705. PMID 2213050
- [Background] Brasil-Neto JP, Pascual-Leone A, Valls-Sole J, Cohen LG, Hallett M. Focal transcranial magnetic stimulation and response bias in a forced-choice task. J Neurol Neurosurg Psychiatry. 1992 Oct;55(10):964-6. doi: 10.1136/jnnp.55.10.964. PMID 1431962